CLINICAL TRIAL: NCT03215693
Title: A Phase II, Multicenter, Single-arm Study to Evaluate Safety and Efficacy of X-396 Capsule in Patients With ALK-positive Non-small Cell Lung Cancer Previously Treated With Crizotinib
Brief Title: X-396 Capsule in Patients With ALK-positive Non-small Cell Lung Cancer Previously Treated With Crizotinib
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTP-42322
Record Dates: First submitted 2017-07-11; First posted 2017-07-12 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-07

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — ensartinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- X-396 capsule (Experimental): 225mg once daily
  Interventions: Drug: X-396 capsule

INTERVENTIONS:
Drug: X-396 capsule — 225mg once daily
  Other Names: Ensartinib

SUMMARY:
The main purpose of the study is to evaluate safety and efficacy of X-396(Ensartinib) capsule in patients with ALK-positive non-small cell lung cancer previously treated with crizotinib.While exploring the relationship between biomarkers and drug efficacy and safety.

DETAILED DESCRIPTION:
This is a phase II, multicenter, single-arm study in which the safety and efficacy of X-396(Ensartinib) will be assessed in adult Chinese patients with ALK-positive(rearrangement) non-small cell lung cancer previously treated with crizotinib. Approximately 144 patients with locally advanced or metastatic NSCLC which carry ALK -rearrangement will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of metastatic non-small cell lung cancer.
* Evidence of positive ALK.
* Patients must have demonstrated progression during or after crizotinib treatment.
* Age 18 years or older at the time of informed consent.
* Eastern cooperative oncology group performance status (ECOG PS) of 0-2
* Measurable disease by response evaluation criteria in solid tumors (RECIST) version 1.1 (v1.1).
* Asymptomatic CNS metastases do not require the use of steroids or anticonvulsants.
* Willingness and ability to comply with the trial and follow-up procedures.
* Ability to understand the nature of this trial and give written informed consent.

Exclusion Criteria:

* Prior use of ALK TKIs with the exception of crizotinib.
* Patients currently receiving cancer system therapy.
* Use of an investigational drug within 4 weeks prior to the first dose of study drug.
* Presence of active gastrointestinal (GI) disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of study medications.
* Patients with a known allergy or delayed hypersensitivity reaction to drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2017-09-28 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) based on independent radiology review | 24 months
  ORR per RECIST 1.1 calculated as the proportion of patients with a best overall response defined as complete response (CR) or partial response (PR).

SECONDARY OUTCOMES:
ORR based on investigator assessment | 24 months
  ORR per RECIST 1.1 calculated as the proportion of patients with a best overall response defined as complete response (CR) or partial response (PR).
Progression-free survival (PFS) as assessed by independent radiology review and investigator | 36 months
  PFS, defined as time from first dose of X-396 to progression or death due to any cause.
Overall survival (OS) | 36 months
  OS, defined as time from first dose of X-396 to death due to any cause.

OTHER OUTCOMES:
Overall intracranial response rate (OIRR) by independent radiology review and investigator assessment | 24 months
  OIRR calculated as the ORR (CR+PR) of lesions in the brain for patients who have measureable disease in the brain at baseline.
Patient reported time to deterioration (TTD) as measured by EORTC C30/LC13 QoL questionnaire | 24 months
  Time to deterioration (TTD) is defined at the time from date of randomization to a worsening of at least 10 points (on a 100 point scale) in each item score of the EORTC C30/LC13

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, MD, Study Chair — Sun Yat-sen University
Locations (4):
- China (4):
  - Beijing Cancer Hospital, Beijing
  - Beijing Chest Hospital，Capital Medical University, Beijing
  - Department of Medical Oncology, Cancer Institute/Hospital, Chinese Academy of Medical Sciences, Beijing
  - Peking Union College Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang Y, Zhou J, Zhou J, Feng J, Zhuang W, Chen J, Zhao J, Zhong W, Zhao Y, Zhang Y, Song Y, Hu Y, Yu Z, Gong Y, Chen Y, Ye F, Zhang S, Cao L, Fan Y, Wu G, Guo Y, Zhou C, Ma K, Fang J, Feng W, Liu Y, Zheng Z, Li G, Wu N, Song W, Liu X, Zhao S, Ding L, Mao L, Selvaggi G, Yuan X, Fu Y, Wang T, Xiao S, Zhang L. Efficacy, safety, and biomarker analysis of ensartinib in crizotinib-resistant, ALK-positive non-small-cell lung cancer: a multicentre, phase 2 trial. Lancet Respir Med. 2020 Jan;8(1):45-53. doi: 10.1016/S2213-2600(19)30252-8. Epub 2019 Oct 15. PMID 31628085